CLINICAL TRIAL: NCT00459914
Title: Sleep Apnea in Patients With Refractory Hypertension: Study of the Prevalence and the Effect of CPAP Treatment on Blood Pressure Control, Endothelial Dysfunction and Angiogenesis.
Brief Title: Sleep Apnea and Refractory Hypertension: Prevalence and Effect of CPAP Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacio Catalana de Pneumologia (Other)
Responsible Party: Ferran Morell, Fundacio Catalana de Pneumologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FUCAP2004
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Hypertension; Sleep Apnea
Keywords: sleep apnea; refractory hypertension; continuous positive airway pressure
MeSH Terms: conditions — Hypertension; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 CPAP (Active Comparator): Nasal continuous positive airway pressure
  Interventions: Device: cpap treatment during sleep
- 2 (No Intervention): Pharmacological treatment alone

INTERVENTIONS:
Device: cpap treatment during sleep — CPAP
  Arms: 1 CPAP

SUMMARY:
A small number of uncontrolled studies have shown a high prevalence of sleep apnea in patients with refractory hypertension and that CPAP treatment achieves a significant reduction of blood pressure in the short term.

The purpose of this study is to assess the prevalence of sleep apnea in patients with refractory hypertension, and the effects of continuous positive pressure treatment on systemic blood pressure and on serum markers of endothelial dysfunction and angiogenesis.

DETAILED DESCRIPTION:
We assess the prevalence of an apnea hypopnea index (AHI) > 5 in patients with refractory hypertension referred from a hypertension clinic. Patients with an AHI >15 are randomized to either continuing their usual pharmacological treatment alone or adding CPAP to their usual treatment, during a 3 month period.

The main endpoint is the comparison of the mean 24h systolic and diastolic blood pressure, as assessed by ambulatory blood pressure monitoring, between both treatment arms. The secondary endpoint is to assess changes in serum markers of endothelial dysfunction and angiogenesis

ELIGIBILITY:
Inclusion Criteria:

* Patients referred from a tertiary hospital hypertension clinic with a diagnosis of refractory hypertension on the basis of office blood pressure higher then 160/90 mmHg despite the recommended doses of at least 3 drugs, including a diuretic.

Exclusion Criteria:

* Causes of secondary hypertension, history of alcohol abuse , renal insufficiency, severe chronically illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-01; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Effect of 3 months of CPAP versus conventional pharmacological treatment on the mean 24 h systolic and diastolic blood pressure . | 3 months

SECONDARY OUTCOMES:
Effect of CPAP versus conventional pharmacological treatment on inflammatory, endothelial function and angiogenesis serum biomarkers | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Lozano, MD, Principal Investigator — Hospital General Universitari Vall d'Hebron; Jose Luis Tovar, MD, Study Chair — Hospital General Universitari Vall d'Hebron; Gabriel Sampol, MD, Study Chair — Hospital General Universitari Vall d'Hebron; Odile Romero, MD, Study Chair — Hospital General Universitari Vall d'Hebron; Pilar Chacon, MD, Study Chair — Hospital General Universitari Vall d'Hebron; Jose Rios, Study Chair — Universitat Autonoma de Barcelona
Locations (1):
- Servei de Pneumologia, Hosital general Universitari Vall d'Hebron, Barcelona, Barcelona, Spain